CLINICAL TRIAL: NCT05586607
Title: Causes and Management of Aseptic Meningitis : A Retrospective Cohort Study in Strasbourg University Hospital
Acronym: Meningitis
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8219
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Aseptic Meningitis
Keywords: Aseptic Meningitis; Infectious; Inflammatory; Neoplastic; Drug-induced
MeSH Terms: conditions — Meningitis, Aseptic; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnostic and therapeutic management of patients with aseptic meningitis is a challenge for the practitioner. There are many etiologies of this condition (infectious, inflammatory, neoplastic, drug-induced), which it is necessary to know how to evoke and look for specifically.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject with aseptic meningitis (CSF pleocytosis, negative bacteriology) from January 2015 to October 2020, at HUS
* Subject having not expressed, after being informed, their opposition to the reuse of their data for the purposes of this research.

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Subject under guardianship or curatorship
* Subject under safeguard of justice
* Positive VZV, HSV, or Enterovirus PCR in CSF
* CSF analysis performed as part of the assessment of a known pathology
* Traumatic or surgical etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) with aseptic meningitis (CSF pleocytosis, negative bacteriology) from January 2015 to October 2020, at HUS
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Retrospective study of the etiologies of aseptic meningitis infection in Alsace | Files analysed retrospectively from January 01, 2015 to October 31, 2020 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine interne et d'Immunologie Clinique - CHU de Strasbourg - France, Strasbourg, France